CLINICAL TRIAL: NCT03927742
Title: Wearable Device Intervention to Improve Sun Behaviors in Melanoma Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: American Cancer Society, Inc. (Other); Melanoma Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019NTLS079; 133512-RSG-19-014-01-CPPB (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2019-04-15; First posted 2019-04-25 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-12

CONDITIONS: Melanoma (Skin)
Keywords: sun protection; sunburn
MeSH Terms: conditions — Melanoma; Sunburn | interventions — Amyloid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shade and application with UV message activated (Experimental): wearable device (wrist) and associated mobile application; UV sensor exposure display and messaging activated
  Interventions: Behavioral: Shade + app with messaging
- Shade and application without UV messaging (Active Comparator): wearable device (wrist) and associated mobile application; UV sensor exposure display and messaging not activated
  Interventions: Behavioral: Shape + app without messaging

INTERVENTIONS:
Behavioral: Shade + app with messaging — Shade wearable device and application with UV messaging activated
  Arms: Shade and application with UV message activated
Behavioral: Shape + app without messaging — Shade wearable device and application without UV messaging activated
  Arms: Shade and application without UV messaging

SUMMARY:
Over 5 million new cases of skin cancer are diagnosed in the United States each year, more than all other cancers combined. Most of these cases are caused by excess exposure to ultraviolet radiation from the sun and artificial sources such as indoor tanning. Melanoma, approximately 87,000 of the annual skin cancer cases and one of the more deadly skin cancers, is on the rise. Previous research on these individuals suggests that while some change how much time they spend in the sun and adopt ways to protect themselves when in the sun, many do not. In our previous study, we found that 20% of melanoma survivors reported a sunburn in the past year and 10% intentionally went outside for a tan, both strong indicators of inappropriate sun exposure. Melanoma survivors are at high risk of second melanomas, making it critical that they spend less time in the sun or take actions to protect themselves when they are in the sun.

No studies to date have investigated technology-based strategies in melanoma survivors to improve sun exposure and protection behaviors. This project will test whether a wearable device that tracks sun exposure and provides alerts regarding sun exposure and protection behaviors will increase sun protection behaviors in melanoma survivors. The use of wearable technology devices (e.g., Fitbit) has grown quickly over the last decade and studies using these devices to promote physical activity and weight loss have been promising. We will test the technology device versus a similar control device in 368 melanoma survivors and compare sun protection behaviors between the two groups.

This project has the potential to identify a strategy that could significantly lower the number of melanoma survivors who go on to have a second melanoma diagnosis. Importantly, this easy to use technology could also be utilized by survivors' family members, who are also at higher risk for melanoma, and the general population as a means to reduce risk of all forms of skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Diagnosed with cutaneous invasive melanoma within HealthPartners system
* Able to read/write in English
* Own a smartphone
* Able to provide voluntary informed consent

Exclusion Criteria:

* Patients who have opted out of their records being used for research purposes
* Inability to provide informed written consent
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogel RI, Luo X, Brown K, Jewett P, Dona AC, Nagler RH, Ahmed RL, Martinson BC, Lazovich D. A UVR-sensor wearable device intervention to reduce sun exposure in melanoma survivors: Results from a randomized controlled trial. PLoS One. 2023 Feb 10;18(2):e0281480. doi: 10.1371/journal.pone.0281480. eCollection 2023. PMID 36763627
- [Derived] Vogel RI, Nagler RH, Ahmed RL, Brown K, Luo X, Martinson BC, Lazovich D. UVR-sensor wearable device intervention to improve sun behaviors and reduce sunburns in melanoma survivors: study protocol of a parallel-group randomized controlled trial. Trials. 2020 Nov 23;21(1):959. doi: 10.1186/s13063-020-04881-3. PMID 33228807

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shade and Application With UV Message Activated | Shade and Application Without UV Messaging
Started | 182 | 186
Completed | 166 | 174
Not Completed | 16 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shade and Application With UV Message Activated | Shade and Application Without UV Messaging | Total
Number analyzed (Participants) | 182 | 186 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.9) | 55.3 (11.5) | 56 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 110 | 221
  Male | 71 | 76 | 147
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 174 | 171 | 345
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 15 | 21

OUTCOME MEASURES:

1. Primary Outcome: Sun Protection Habits Index
Description: Sun protection habits measured using Glanz et al., 2008 questionnaire and scored by taking the averaging of 6 protective behaviors (wearing a shirt with sleeves, wearing sunglasses, staying in the shade, using sunscreen, limiting time in the sun, and wearing a hat) on a 4-point ordinal scale ranging from 1 = rarely or never to 4 = always. (Glanz et al. 2010).
  Higher score indicates better sun protection behaviors
Time Frame: 12 weeks (post intervention)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Shade and Application With UV Message Activated | Shade and Application Without UV Messaging
Number analyzed (Participants) | 166 | 174
scores on a scale | 2.9 (0.5) | 3 (0.5)

2. Secondary Outcome: Number of Participants With Sunburn in the Past 12 Weeks
Description: Glanz et al. (2007) validated question: In the past 12 months, how many times did you have a red OR painful sunburn that lasted a day or more? Self-reported options include 0, 1, 2, 3, 4, 5 or more.
Time Frame: 12 weeks (post intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Shade and Application With UV Message Activated | Shade and Application Without UV Messaging
Number analyzed (Participants) | 166 | 174
Participants | 55 | 54

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Shade and Application With UV Message Activated | Shade and Application Without UV Messaging
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/174
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/174
Other Adverse Events (participants affected / at risk) | 0/166 | 0/174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03927742/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03927742/ICF_001.pdf